CLINICAL TRIAL: NCT05736380
Title: The Effects of Cerebellar rTMS on Brain Activity
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Requires funding to commence fMRI scan - funding awaited
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Prof Shaheen Hamdy PhD FRCP, Professor, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRAS 256390
Record Dates: First submitted 2022-11-30; First posted 2023-02-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: The Effects of Cerebellar rTMS on the Brain

STUDY DESIGN:
Intervention Model Description: Over the course of two visits to the laboratory, each participant will undergo either real or sham cerebellar rTMS. Afterwards they will have functional magnetic resonance imaging of their brains.
Who Masked: Participant
Masking Description: Over the course of two visits to the laboratory, each participant will be randomised to either real or sham cerebellar rTMS. Each participant will undergo both procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral cerebellar rTMS (Active Comparator)
  Interventions: Device: Cerebellar rTMS
- Sham cerebellar rTMS (Sham Comparator)
  Interventions: Device: Sham cerebellar rTMS

INTERVENTIONS:
Device: Cerebellar rTMS — 250 pulses at 10 Hertz over the cerebellum
  Arms: Unilateral cerebellar rTMS
Device: Sham cerebellar rTMS — Sham cerebellar rTMS
  Arms: Sham cerebellar rTMS

SUMMARY:
Swallowing function is controlled by two swallowing centres (one on each half of the brain). There is a dominant and non-dominant swallowing centre. Damage to any part of the brain can lead to swallowing problems, for example in strokes. Recovery of the ability to swallow is associated with increased activity (compensation) over the undamaged centre. The cerebellum is an area of the brain involved in the control and modulation of muscle movements. It is found at the back of the skull. Anatomical evidence exists, showing cerebellar outputs projecting to several cortical areas, including the primary motor cortex (M1). Moreover, brain imaging studies have shown activation of the cerebellum during swallowing using positron emission tomography (PET) and magnetic resonance imaging (MRI).

Over the past few years studies have tried to improve swallowing function using techniques to stimulate regions of the brain and encourage compensation. Repetitive transcranial magnetic stimulation (rTMS) is a technique which can temporarily increase or suppress activity over regions of the brain. No imaging studies have been conducted which have looked at how the brain is affected by cerebellar rTMS.

The investigators hypothesise that cerebellar rTMS will cause increased activity in swallowing associated areas in the brain, including the cortex and brainstem

DETAILED DESCRIPTION:
Experiment The optimal motor stimulation sites for pharyngeal and thenar cortical areas and the cerebellum will be identified and marked using single pulse TMS with a coil. Anatomical landmarks will be used to help guide neuronavigation. The vertex (top) of the head will be identified with a tape measure as will the inion (the most prominent part at the back of the skull). Studies have demonstrated that pharyngeal (throat) and thenar (thumb) cortical areas are found in front and to the side of the vertex while both halves of the cerebellum lie below and to the side of the inion. The thenar resting motor threshold over the dominant pharyngeal hemisphere is required for calculation of cerebellar rTMS intensity.

Participants will then be randomly allocated to either real right sided cerebellar rTMS or sham (pretend) cerebellar rTMS on each visit. Each participant will undergo both procedures (real and sham) over the course of their involvement with the study. Real cerebellar rTMS will be delivered by holding the figure of eight coil flat against the head. It will be administered at 90% of thenar resting motor threshold at a frequency of 10 Hertz. Sham cerebellar rTMS will be delivered by holding the coil perpendicular to the scalp with only the edge of the coils making contact with the head. This technique has been used in previous studies and will ensure that no stimulation is delivered to the cerebellum.

After real or sham cerebellar rTMS, participants will have functional magnetic resonance imaging (fMRI) scans of their brains. During the scan participants will be asked to swallow water through a plastic tube. This will activate their brain swallowing centres. Each participant will be asked to complete five swallowing cycles. Each cycle will involve swallowing 10 times with a one second gap between swallows. Cycles will be separated by a 10 second period of rest.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults above 18 years of age

Exclusion Criteria:

1. Epilepsy
2. Cardiac pacemaker
3. Previous brain surgery
4. Previous swallowing problems
5. The use of medication which acts on the central nervous system
6. Any implanted metal in the head

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Differential blood flood (fMRI) | 15 minutes post cerebellar rTMS
  Differential blood flow in brain regions post cerebellar rTMS (compared to sham)

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Hamdy, Principal Investigator — University of Manchester
Locations (1):
- Upper G.I laboratory, Salford Royal Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No